CLINICAL TRIAL: NCT00019201
Title: PILOT STUDY OF THE CORRELATION BETWEEN THE FINDINGS OF ATYPICAL/MALIGNANT CELLS IN SPUTUM AND FLUORESCENCE BRONCHOSCOPY IN PATIENTS AT RISK FOR LUNG CANCER OF THE LIFE IMAGING SYSTEM AND WHITE LIGHT BRONCHOSCOPY
Brief Title: Fluorescent Light Bronchoscopy Plus White Light Bronchoscopy for Early Detection of Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Screening
Other Study IDs: CDR0000065062; NCI-96-C-0128; NCT00001511 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2000-02

CONDITIONS: Head and Neck Cancer; Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage III non-small cell lung cancer; limited stage small cell lung cancer; stage I nasopharyngeal cancer; stage II nasopharyngeal cancer; stage III nasopharyngeal cancer; stage I lip and oral cavity cancer; stage II lip and oral cavity cancer; stage III lip and oral cavity cancer; stage I hypopharyngeal cancer; stage II hypopharyngeal cancer; stage III hypopharyngeal cancer; stage I laryngeal cancer; stage II laryngeal cancer; stage III laryngeal cancer; stage I paranasal sinus and nasal cavity cancer; stage II paranasal sinus and nasal cavity cancer; stage III paranasal sinus and nasal cavity cancer; stage I oropharyngeal cancer; stage II oropharyngeal cancer; stage III oropharyngeal cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Nasopharyngeal Neoplasms; Mouth Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Oropharyngeal Neoplasms | interventions — Immunohistochemistry; Bronchoscopy; Endoscopic Mucosal Resection

INTERVENTIONS:
Other: cytology specimen collection procedure
Other: immunohistochemistry staining method
Other: sputum cytology
Procedure: bronchoscopic and lung imaging studies
Procedure: bronchoscopy
Procedure: comparison of screening methods
Procedure: endoscopic biopsy

SUMMARY:
RATIONALE: Fluorescent bronchoscopy, when used in combination with conventional white light bronchoscopy, may improve the ability to detect early lung cancer.

PURPOSE: A pilot study to evaluate fluorescent light bronchoscopy plus conventional bronchoscopy as a tool for screening and detecting lung cancer in persons with completely resected head and neck cancer or successfully treated early-stage lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the efficacy of autofluorescence bronchoscopy using the Lung Imaging Fluorescence Endoscopic System with conventional white-light bronchoscopy for the early detection of lung cancer in selected patients with known or suspected bronchogenic carcinoma, completely resected head and neck cancer, and successfully treated early-stage lung cancer.
* Determine the number of areas of moderate dysplasia, severe dysplasia, and carcinoma in situ in patients treated with surgery for lung cancer compared with patients treated with combined modality therapy.
* Determine the ability of immunohistochemistry to predict whether lesions of moderate to severe dysplasia will progress to cancer.

OUTLINE: If possible, patients produce a 3-day pooled sputum sample prior to bronchoscopy. Patients then undergo tracheobronchial white-light bronchoscopy followed by autofluorescence bronchoscopy using the Lung Imaging Fluorescence Endoscopic (LIFE) Device attached to a computerized video camera. Visualized tissue is classified as either normal, abnormal, or suspicious. Abnormal or suspicious tissue is biopsied, as is tissue from 1 or 2 randomly chosen normal sites. Immunohistochemical analysis of the biopsy material is conducted without knowledge of the bronchoscopic results. Patients unable to produce a sputum sample prior to bronchoscopy are required to do so after bronchoscopy.

PROJECTED ACCRUAL: A total of 70 patients will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* The following diagnoses are eligible:

  * Known or suspected bronchogenic carcinoma scheduled for bronchoscopy as part of standard diagnostic or staging work-up
  * Completely resected stage I/II non-small cell lung cancer with no evidence of metastasis
  * Stage III non-small cell lung cancer with no evidence of disease for at least 2 years following treatment
  * Small cell lung cancer with no evidence of disease for at least 2 years following treatment
  * Completely resected head and neck cancer with no evidence of metastasis
* Ability to produce sputum samples required

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Hematopoietic:

* WBC 2,000-20,000
* Platelets at least 50,000

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No uncontrolled hypertension (i.e., systolic pressure greater than 200 mm Hg or diastolic pressure greater than 120 mm Hg)
* No unstable angina

Other:

* No bleeding disorder
* No allergic reaction to topical lidocaine
* No pregnant women

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* At least 18 months since ionizing radiotherapy to the chest

Surgery

* See Disease Characteristics

Other

* At least 1 month since yttrium-aluminum-garnet (YAG) laser therapy to the lung
* At least 3 months since fluorescent photosensitizing drugs (e.g., Photofrin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-08

CONTACTS AND LOCATIONS:
Overall Officials: J. Michael Hamilton, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States